CLINICAL TRIAL: NCT05807841
Title: Influence of Novel Intravascular Ultrasound-Based Artificial Intelligence Technologies on Event Reduction Following Percutaneous Coronary Intervention (INNOVATE-PCI)
Brief Title: Clinical Impact of Intravascular Ultrasound-Based Artificial Intelligence Technologies (INNOVATE-PCI)
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Seung-Whan Lee, M.D., Ph.D., Principal Investigator, Asan Medical Center
Other Study IDs: 2020-0226
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease
Keywords: percutaneous coronary intervention; artificial intelligence; machine learning; intravascular ultrasound; coronary angiography
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: percutaneous coronary intervention — IVUS-guided stent implantation

SUMMARY:
This study is a prospective, multicenter study in the real practice to validate the diagnostic performances and clinical impact of coronary angiography & intravascular ultrasound (IVUS)-based models developed by machine learning (ML).

DETAILED DESCRIPTION:
The aim of the study is to evaluate the performances and prognostic impact of coronary angiography & IVUS-based algorithms for decision making and stent optimization in a multicenter, prospective cohort. Between January 2020 and June 2025, a total of 3,000 patients who performed coronary angiography (± FFR) and have at least one coronary stenosis requiring PCI (as culprit) will be enrolled from 15 centers in South Korea. In addition, the deferred lesions with visual estimated diameter stenosis of >30% will be evaluated as non-culprits. Brief study design is as depicted in the following figure.

Supervised ML algorithms include: 1) angiography- and IVUS-based algorithms for predicting FFR, 2) IVUS-based algorithm for plaque characterization, 3) IVUS-based algorithm for predicting stent expansion, and 4) post-stenting IVUS-based algorithm for predicting stent failure. In the prospective cohort, the performance of each model will be assessed. This registry trial composed of the treated (culprit) and the deferred (nonculprit) coronary lesions has two primary objectives as follow; 1) Primary objectives in treated (culprit) lesions is to see the impact of the integrated ML model on the development of culprit-related 2-year target vessel failure (TVF). 2) Primary objectives in deferred (nonculprit) lesions is to see the impact of the integrated ML model on the development of nonculprit-related 2-year TVF.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Symptomatic angina patients with objective myocardial ischemia
* Patients with at least one major epicardial coronary artery that requires stent implantation
* Subject who signs with informed consent form

Patient exclusion Criteria:

* ST-segment elevation MI at admission
* Patients who underwent coronary artery bypass surgery or heart transplantation
* Left ventricular ejection fraction <30%
* Cardiogenic shock
* Patients whose life expectancy <2 years
* Woman who are breastfeeding, pregnant or planning to become pregnant during study
* Patients in whom anti-platelets or heparin is contraindicated

Lesion exclusion Criteria:

* Left main culprit lesion (angiographic diameter stenosis >50%)
* Thrombus-containing lesion
* In-stent restenosis
* Side branch lesion
* Chronic total occlusion
* Small vessel with reference diameter <2.5mm
* Coronary spasm despite administration of nitrate
* Inability for imaging catheter to pass through tight stenosis, calcification, angulations
* Poor image quality
* Angiographically visible collateral vessels

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between February 2020 and June 2025, a total of 3,000 patients who performe coronary angiography (± FFR) and have at least one coronary stenosis requiring PCI (as culprit) will be enrolled from 15 centers in South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
culprit-related TVF | 2 years after stent implantation
  composite of cardiac death, myocardial infarction (MI), stent thrombosis, and clinically-driven target vessel revascularization (TVR) at 2 years after SynergyTM implantation
nonculprit-related TVF | 2 years after stent implantation
  composite of cardiac death, MI, and clinically-driven TVR at 2 years

SECONDARY OUTCOMES:
each component of primary measures | 2 years after stent implantation
  each of cardiac death, non-fetal MI, ST and target vessel revascularization
all cause death | 2 years after stent implantation
  all cause death
repeat revascularization | 2 years after stent implantation
  repeat revascularization
stroke | 2 years after stent implantation
  stroke
bleeding | 2 years after stent implantation
  bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Whan Lee, MD, Principal Investigator — Asan Medical Center
Locations (16):
- South Korea (16):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Gosin University Gospel Hospital, Busan
  - Inje University Pusan Paik Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Kangwon National University Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic university of korea, daejeon st. mary's hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Jesushospital, Jeonju
  - Chungnam National University Sejong Hospital, Sejong
  - Seung-Whan Lee, Seoul
  - Kangbuk Samsung Medical Center, Seoul
  - The Catholic university of korea, Eunpyeong st. mary's hospital, Seoul
  - Veterans Hospital Service Medical Center, Seoul
  - The Catholic University of Korea ST.VINCENT'S Hospital, Suwon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: Undecided